CLINICAL TRIAL: NCT04864366
Title: Efficacy and Safety of TAF for 48 Weeks in HBeAg Positive CHB Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, chief physician,professor, Huashan Hospital
Other Study IDs: TAF-HBeAg-CHB
Record Dates: First submitted 2021-04-09; First posted 2021-04-28 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment naive patients: 1. HBV DNA> 20000 IU/ml
  2. ALT>2×ULN；or ALT>1×ULN，but liver biopsy showed inflammation greater than or equal to G2, or/and liver fibrosis greater than or equal to S2
  3. No treatment with NA or/or αIFN within 1 year
  Interventions: Drug: Tenofovir Alafenamide 25 MG [Vemlidy]
- ETV treatment experienced patients: 1. ETV treatment for 1 to 2 years before
  2. HBsAg>3000IU/mL
  3. HBV DNA<20IU/mL
  4. ALT<1×ULN
  5. No other NA therapy prior to entecavir treatment
  6. Patients had a desire to convert to TAF therapy
  Interventions: Drug: Tenofovir Alafenamide 25 MG [Vemlidy]

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG [Vemlidy] — TAF is administered as a 25mg/tablet, taken orally with food once daily, for 48 weeks.

SUMMARY:
The objective of this clinical study was to observe the changes of HBsAg levels after a sequential 48 weeks-treatment of TAF in ETV experienced CHB patients and to monitor the levels of cytokines such as IFN-λ3, IP-10, IL-12, IL-10, and IL-21.

DETAILED DESCRIPTION:
The first-line NAs include entecavir (ETV), tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF). All the NAs mentioned above could achieve complete virologic response. NAs mentioned above are sufficient in inhibiting viral replication. However, there may exist difference in long-term prognosis such as HBsAg level decline, resistance development and HCC development. A prospective study performed by our team previously showed that TDF was better than ETV in HBsAg decline. A Korean research showed that TDF therapy was associated with a significantly lower risk of HCC than ETV therapy; the TDF group showed a distinct reduction in HBsAg level after one-year treatment. Also, a Japanese RCT study indicated that the reduction in HBsAg level was significantly greater in the TDF arm than the ETV arm at week 24. The mechanism of HBsAg decline induced by TDF has not been fully elucidated. Patients treated with nucleotide analogues (adefovir, tenofovir) had higher serum IFN-λ3 levels than those treated with nucleoside analogues (lamivudine, entecavir), according to results recently published in Gut. A team from Japan has found that nucleotide analogues inhibit LPS-mediated IL-10 production and induce IL-12p70 and TNF-α production. We speculated that, compared with entecavir, tenofovir could up-regulate IFN-λ3 and reduce the level of HBsAg more significantly.

As known as the second generation of TDF, TAF has a significantly longer half-life than TDF. A phase 3 study displayed that TAF 25 mg was non-inferior to TDF 300 mg in suppressing HBV replication, with a better performance in renal and bone safety. However, there is lack of study evaluating TAF in reducing HBsAg and induces IFN-λ3.The aim of this study was to investigate whether the TAF can achieve a better antiviral therapeutic endpoint, i.e. a greater reduction in HBsAg levels, or even meet the therapeutic expectation of stopping NAS in a larger number of treated patients.

The objective of this clinical study was to observe the changes of HBsAg levels after a sequential 48 weeks-treatment of TAF in ETV experienced CHB patients and to monitor the levels of cytokines such as IFN-λ3, IP-10, IL-12, IL-10, and IL-21.

ELIGIBILITY:
common criteria:

* Age 18-70 years old (including both ends), male or female, chronic HBV infection (HBsAg positive for more than 6 months, or liver biopsy results show chronic hepatitis B infection)
* HBsAg positive
* Patient must be capable of understanding and signing written informed consent; Before commencing the study procedure, participants must obtain informed consent.
* Lifestyle requirements:

All subjects considered by the investigator to be sexually active and capable of becoming pregnant or making sexual partner become pregnant must agree to use an effective contraceptive method for the entire study period (from the signing of the informed consent to at least 28 days after the last dose of the investigational drug was administered).

Addition criteria:

Treatment naive patients

* HBV DNA> 2×104 IU/ml
* ALT>2×ULN；or ALT>1×ULN，but liver biopsy showed inflammation greater than or equal to G2, or/and liver fibrosis greater than or equal to S2
* No treatment with NA or/or αIFN within 1 year

ETV treatment experienced patients

* ETV treatment for 1 to 2 years before
* HBsAg>3000IU/mL
* HBV DNA<20IU/mL
* ALT<1×ULN
* No other NA therapy prior to entecavir treatment
* Patients had a desire to convert to TAF therapy

Exclusion Criteria:

Treatment naive patients

* treated with NA or/or αIFN within 1 year
* Pregnant women, lactating women, or women who plan to become pregnant within 2 years
* Co-infection with Hepatitis C, Hepatitis D or HIV;
* Chronic liver diseases with non-HBV etiology (including but not limited to: autoimmune hepatitis, primary biliary cirrhosis, primary cirrhosis cholangitis, hemochromatosis, etc.
* There is evidence of Child-Pugh grade C decompensated liver disease, or moderate to severe ascites, and grade III-IV hepatic encephalopathy
* There are symptoms and signs of hepatocellular carcinoma. If screening for alpha-fetoprotein (AFP) <50 ng / mL, imaging examination are not required; but if screening for AFP> 50 ng / mL, imaging examination are required
* current alcohol or drug abuse may affect compliance
* Patients who recieved solid organ or bone marrow transplantation. Liver or kidney transplantation patients can be enrolled
* malignant tumors within 5 years. Patients being evaluated for possible malignant tumors should be excluded
* Study drugs were used within 3 months prior to screening
* Patients who are participating in other clinical trials, or have been treated with the study drugs within 12 weeks before screening
* Inability or unwillingness to provide informed consent or non-compliance with research requirements
* Patients who are unwilling to purchase TAF on their own
* In addition to the above exclusion criteria, patients who meet any of the contraindications listed in the label of the investigational drug product

ETV treatment experienced patients

●Patients who had received IFN and/or other NA (except entecavir) within 1 year Other exclusion criteria were as same as 2-13 of the exclusion criteria for treatment naive patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-positive men, non-pregnant women and non-lactating women (over 18 years of age) who are infected with HBV alone, treatment naïve or only ETV treatment experienced at least 48 weeks. participate will only receive TAF treatment after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-10-27 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum HBsAg at week 48 from baseline. | from baseline to week 48 after TAF treatment
  evaluate the changes of serum HBsAg level after 48 week-treatment of TAF in TN and ETV experienced CHB patients.

SECONDARY OUTCOMES:
Change of serum HBeAg level from baseline. | from baseline to week 48 after TAF treatment
  evaluate the of changes serum HBeAg level from baseline after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of serum HBcAb level from baseline. | from baseline to week 48 after TAF treatment
  evaluate the of changes serum HBcAb level from baseline after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
propotion of patients who maintened HBV DNA suppression. | from baseline to week 48 after TAF treatment
  evaluate the propotion of patients who maintened HBV DNA suppression after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
propotion of patients who maintened ALT normalization. | from baseline to week 48 after TAF treatment
  evaluate the propotion of patients who maintened ALT normalization after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers - eGFR from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers -eGFR after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers - serum phosphate from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers -serum phosphate after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers - UPCR from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers - UPCR after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers- UACR from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers - UACR after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers - RBP:Cr from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers -RBP:Cr after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of renal markers - β2MG:Cr from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of renal markers - β2MG:Cr after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of IFN-λ3 from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of IFN-λ3 after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of IP-10 from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of IP-10 after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of IL-12 from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of IL-12 after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of IL-10 from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of IL-10 after 48 week-treatment of TAF in TN and ETV experienced CHB patients.
Change of IL-21from baseline. | from baseline to week 48 after TAF treatment
  evaluate the change of IL-21 after 48 week-treatment of TAF in TN and ETV experienced CHB patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jiming Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (3):
- China (3):
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Ruijin Hospital Affiliate to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai